CLINICAL TRIAL: NCT02301221
Title: A Study of Efficacy, Safety and Durability of Fecal Microbiota Transplantation in Adult Patients With Slow Transit Constipation
Brief Title: Effect of Fecal Microbiota Transplantation in Slow Transit Constipation
Acronym: FMTSTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinling Hospital, China (Other)
Responsible Party: Principal Investigator, Jianfeng Gong, Associate professor, Jinling Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIGS-FMT-STC-2014
Record Dates: First submitted 2014-11-11; First posted 2014-11-25 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Slow Transit Constipation
Keywords: Fecal Microbiota Transplantation; Slow Transit Constipation; Colonic motility
MeSH Terms: interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Fecal microbiota transplantation (FMT) (Experimental): Patients included will receive standard FMT, and then will be followed up for 24 weeks.
  Interventions: Procedure: Fecal microbiota transplantation (FMT); Drug: Vancomycin and bowel lavage

INTERVENTIONS:
Procedure: Fecal microbiota transplantation (FMT) — Standardized Frozen Fecal Microbiota will be infused via nasointestinal tube.
  Other Names: Fecal bacteriotherapy
Drug: Vancomycin and bowel lavage — An initial vancomycin regimen (500 mg orally two times per day for 3 days), followed by bowel lavage before the infusion of a solution of donor fecal microbiota.

SUMMARY:
The purpose of this study is to evaluate the effect of fecal microbiota transplantation in adults with slow transit constipation.

DETAILED DESCRIPTION:
Constipation is a chronic disease estimated to affect about 10% - 15% of the worldwide general population. Constipation frequency appears to augment with increasing age, particularly after 65 years old.

Recent evidence in the literature and collected in our laboratory confirm that constipation can be a consequence of intestinal dysbiosis, with an increase of potentially pathogenic microorganisms and a decrease of potentially beneficial microorganisms. These alterations may affect the motility and metabolic environment of colon, especially the production of short chain fatty acids (SCFAs).

A new and under-explored method to manipulate the gastrointestinal microbiota involves fecal microbiota transplantation (FMT). There has been growing interest in the use of fecal microbiota for the treatment of patients with chronic gastrointestinal infections (e.g. CDI) and other extraintestinal conditions (e.g. IBD). Similarly, we suppose that reshaping the gut microbiome with FMT would be effective for patients with slow transit constipation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic constipation according to Rome III criteria, defined as two or fewer spontaneous, complete bowel movements (SCBMs) per week for a minimum of 6 months;
* Age ≥ 18 years;
* BMI: 18.5-25 kg/m2;
* Slow colonic transit confirmed by colonic transit test (colonic transit time (CTT) > 48 hours);
* Normal anorectal manometry with no evidence of dyssynergia and confirmed ability to expel rectal balloon;
* No radiographic evidence of functional (i.e. pelvic floor dyssynergia) or anatomical (i.e. significant rectocele and intussusception) impediment to the expulsion of the radio-opaque contrast;
* Disease duration > 1 year;
* Traditional treatment with dietary modification, laxatives (including osmotic and stimulant laxatives), and biofeedback tried over the past 6 months without success;

Exclusion Criteria:

* Bowel constipation due to innate factor (i.e. megacolon) or secondary interventions (i.e. drugs, endocrine, metabolic, neurologic or psychologic disorders);
* History or evidence of gastrointestinal diseases (i.e. obstruction, cancer, inflammatory bowel diseases) ;
* Previous abdominal surgery, except cholecystectomy, appendicectomy, tubal ligation and cesarean section;
* Previous proctological or perianal surgery;
* A constipation condition meeting the Rome III criteria for IBS or functional abdominal pain syndrome;
* Pregnant or breast-feeding women;
* Infection with enteric pathogen;
* Usage of probiotics, prebiotics and/or synbiotics within the last month;
* Usage of antibiotics and/or PPIs within the last 3 months;
* Smoking or alcohol addiction within the last 3 months;
* Uncontrolled hepatic, renal, cardiovascular, respiratory or psychiatric disease;
* Disease or therapy with drugs (i.e. antidepressants, opioid narcotic analgesics, anticholinergics, calcium antagonists, nitrates, antimuscarinics) that, in the opinion of the investigator, could affect intestinal transit and microbiota.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-03 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients having on average three or more SCBMs/week | 24 weeks
  Proportion of patients having on average three or more spontaneous, complete bowel movements (SCBMs) per week was evaluated at baseline and over the week interval 3-4, 9-12 and 21-24.

SECONDARY OUTCOMES:
Bowel habit assessments | 24 weeks
  Patients kept daily diaries about times of bowel movements each day, stool consistency, degree of straining severity during defecation, and degree of sensation of incompleteness of evacuation.
Constipation-related symptoms assessments | 24 weeks
  Constipation-related symptoms were evaluated using the validated Patient Assessment of Constipation Symptoms (PAC-SYM) questionnaire at baseline and at week 4, 12, and 24.
Quality-of-Life assessments | 24 weeks
  Quality-of-Life was evaluated using the validated Patient Assessment of Constipation Quality of Life (PAC-QOL) self-report questionnaire at baseline and at week 4, 12, and 24.
Colonic transit time measurements | 24 weeks
  Colonic transit time (CTT) was measured at baseline and at week 4, 12 and 24 with the Metcalf method.
Usage of laxatives or enemas as rescue medication | 24 weeks
  If patients did not have a bowel movement for 3 or more consecutive days, they were permitted to take up to 20 g of Macrogol 4000 powder (Forlax). If ineffective, enema were used. Patients kept daily diaries about the rescue medication when used.
Adverse events | 24 weeks
  Adverse events include fever, diarrhea, abdominal pain, increased bloating, borborygmi, flatulence, nausea, vomiting, nasopharyngitis, and any other disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, MD, Study Director — Department of Generay Surgery, Jinling hosptal
Locations (1):
- Department of Generay Surgery, Jinling hosptal, Medical School of Nanjing University, Nanjing, Jiangsu, China